CLINICAL TRIAL: NCT01570088
Title: Bioavailability of Folic Acid and L-5-methyltetrahydrofolic Acid in Fortified Bread: a Randomized Placebo-controlled Trial
Brief Title: Bioavailability of Folic Acid Fortified Bread
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: H12-00339
Record Dates: First submitted 2012-03-16; First posted 2012-04-04 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Red Blood Cell Folate
MeSH Terms: interventions — Folic Acid; 5-methyltetrahydrofolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Folic acid (Active Comparator)
  Interventions: Dietary Supplement: Folic acid
- L-5-MTHF (Experimental)
  Interventions: Dietary Supplement: L-5-MTHF
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Folic acid — One roll/bun per day fortified with 400 µg of folic acid
  Arms: Folic acid
Dietary Supplement: L-5-MTHF — One roll/bun per day fortified with 452 µg of L-5-MTHF
  Arms: L-5-MTHF
Other: Placebo — Placebo contains no folic acids
  Arms: Placebo

SUMMARY:
Folic acid is the synthetic form of vitamin folate. Because of its high stability and bioavailability, it is the form of folate added to bread in Canada to reduce birth defects. There are health concerns about long-term folic acid consumption. Another form of folate, L-5-methyltetrahydrofolic acid (L-5-MTHF) has become available which does not have these health concerns. Unfortunately L-5-MTHF is not as stable as folic acid, but the investigators have developed a method to stabilize L-5-MTHF in food. The investigators plan to conduct a randomized trial to compare the bioavailability of bread fortified with L-5-MTHF versus folic acid.

The investigators hypothesize that bread fortified with L-5-MTHF will increase red cell folate over 16 weeks to the same extent as bread fortified with equimolar folic acid.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Not taking a folic acid containing supplement

Exclusion Criteria:

* Adults who have medical conditions such as diabetes, asthma, cancer, cardiovascular disease, high blood pressure, celiac disease, or psychiatric illness
* Adults who are taking medications known to interfere with folate metabolism (i.e. phenytoin, sulphasalazine, methotrexate)
* Adults with wheat, milk allergy or lactose intolerance
* Adults with known B12 deficiency
* Adults who consume more than 1 alcoholic drink/day on average (1 drink=12 oz beer, 5 oz wine or 1.5 oz spirits)
* Women have been pregnant during the year previous
* Women planning a pregnancy in the next year
* Women who believe they may become pregnant during the study
* Women who have had a known previous neural tube defect affected pregnancy
* Adults who are unable to provide informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
red blood cell folate concentration at three time points | baseline, 8th week, 16th week
  We will take one blood sample at baseline, 8th and 16th week. For each blood sample, we will measure the red blood cell folate concentration as our primary outcome measure. We will record the changes in the folate concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Green, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Green TJ, Liu Y, Dadgar S, Li W, Bohni R, Kitts DD. Wheat rolls fortified with microencapsulated L-5-methyltetrahydrofolic acid or equimolar folic acid increase blood folate concentrations to a similar extent in healthy men and women. J Nutr. 2013 Jun;143(6):867-71. doi: 10.3945/jn.113.174268. Epub 2013 Apr 24. PMID 23616513